CLINICAL TRIAL: NCT02284503
Title: A 30-day, Randomized, Open-Label, Multicenter Study Exploring Efficacy of Intensive Rosuvastatin Treatment Peri-PCI in Chinese Patients With NSTE-ACS
Brief Title: Exploring Efficacy of Intensive Rosuvastatin Treatment Peri-PCI in Chinese Patients With Non ST-segment Elevated Acute Coronary Syndrome(NSTE-ACS)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISSCRES0169
Record Dates: First submitted 2014-10-30; First posted 2014-11-06 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-11

CONDITIONS: Non-ST-elevation Acute Coronary Syndromes
Keywords: MI reduction; intensive statin treatment; NSTE-ACS
MeSH Terms: interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 40mg Rosuvastatin group (Experimental): The subjects in this group will receive Rosuvastatin 40mg within 12±2h before PCI, follow 20mg post PCI for 30days.
  Interventions: Drug: Rosuvastatin
- 20mg Rosuvastatin group (Experimental): The subjects in this group will receive Rosuvastatin 20mg within 12±2h before PCI, follow 20mg post PCI for 30days.
  Interventions: Drug: Rosuvastatin
- no statin group (Experimental): The subjects in this group will not receive Rosuvastatin before PCI, follow 10mg post PCI for 30days.
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — The subjects will receive intensive Rosuvastatin before and after PCI
  Other Names: Rosuvastatin Calcium Tablets

SUMMARY:
This is a 30-day, randomized, open-label, 3-arm, parallel-group, multicenter study exploring efficacy of intensive rosuvastatin treatment peri-PCI in Chinese patients with NSTE-ACS.

DETAILED DESCRIPTION:
Non ST-segment elevated acute coronary syndrome(NSTE-ACS) is increasing rapidly, and is more frequent than ST-segment elevated acute coronary syndrome (STE-ACS) now. NSTE-ACS patients sent to early PCI procedure is large and increasing rapidly in China.Quite a few trials have focused on high loading dose statin before PCI to improve cardiovascular outcomes in ACS. In Asian, high loading dose statin therapy showed different outcome. Rosuvastatin (RSV) is one of the most potent statins.Nowadays, quite a few experts think ACS patients undergoing PCI not only need loading dose statin, but also post PCI intensive statin treatment is rather important. Chinese consensus and western guidelines recommend intensive statin treatment in these patients. However, Chinese consensus referred to the western study as there's no relevant intensive statin treatment peri-PCI study in China until now.

Thus this study is designed to explore the efficacy of intensive statin treatment peri-PCI (early loading dose-RSV 40 mg or 20mg before PCI and subsequent 20mg post PCI) in periprocedural myocardial injury and 30 days MACE reduction in Chinese NSTE-ACS patients and explore efficacy of 30-day RSV 20 mg post-PCI treatment in lipid profile, inflammatory factors compared with baseline.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 year old males and non-child-bearing period females.
2. Clinical diagnosed with NSTE-ACS, including unstable angina or non-ST-segment elevation myocardial infarction(NSTEMI).

   * For unstable angina, the diagnose should meet all below:

   Clinical onset features: angina for at least 20 min when resting; initial onset angina pectoris(new onset within one month) manifests spontaneous angina or labor angina (CCS grade II or III); Symptoms of original stable angina pectoris aggravate in one month and at least achieve CCS grade III (accelerated angina pectoris); angina onset within one month after MI.

   ECG: At least twice in one month: ST depression or elevation >0.1millivolt (mv) or T-wave inversion ≥0.2 mv in 2 or more contiguous electrocardiographic leads when onset and the ST-T changes recovered after remission of chest pain. Myocardial damage marker do not elevate or reach the MI diagnostic level.
   * For NSTEMI, the diagnose should meet all below ischemia symptoms(ischemic chest pain lasting more than 30 min and cannot relief significantly by sub-lingual NTG) ECG change: new ST-T dynamic development (new or transient ST depression ≥0.1mv or T-wave inversion≥0.2mv).

   Myocardial damage marker level is normal or elevated to the MI diagnostic level.
3. Received early (within 48 h) Percutaneous Coronary Intervention(PCI).
4. Should be statin- naïve(last 3 months).
5. Only receive drug-eluting stents.
6. Sign the Informed Consent Form(ICF)

Exclusion Criteria:

Any of the following is regarded as a criterion for exclusion from the study:

1. Diagnosis as STEMI;
2. NSTE-ACS with high-risk features warranting emergency coronary angiography;
3. Receive only medical therapy or Coronary Artery Bypass Graft(CABG)
4. Active liver disease or dysfunction including agnogenic serum transaminase sustained elevation or higher than 3 times upper limit of normal(ULN);
5. Left ventricular ejection fraction<30%;
6. Previous or current treatment with statins;
7. Patients with myopathy or serum creatine kinase > 5 times the upper limit of normal not caused by myocardial injury;
8. Severe renal function damage (creatinine clearance rate<30 ml/min);
9. Severe anemia (haemoglobin< 6g/L);
10. Diagnosed with malignancy within 5 years;
11. Concurrent use ciclosporin；
12. Investigator evaluated as not appropriate for statins.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1350 (Estimated)
Dates: Start 2014-11; Primary Completion 2014-12 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
myocardial injury reduction | 30 days
  Myocardial injury assessed by creatine kinase-MB. (CK-MB) elevation, defined as a post-procedural elevation of CK-MB values >3×99th percentile Upper Reference Limit (URL) in patients with normal baseline values >99th percentile URL or a rise of CK-MB values>20% if the baseline values are elevated and are stable or falling; or assessed by cTn elevation, defined as a post-procedural elevation of cardiac troponin (cTn) values >5×99th percentile URL in patients with normal baseline values >99th percentile URL or a rise of cTn values>20% if the baseline values are elevated and are stable or falling.

SECONDARY OUTCOMES:
MACE reduction | 30 days
  Major Adverse Cardiac Events(MACE) event including death, Myocardial infarction(MI), target vessel revascularization, ischemic stroke
the change of lipid | 30 days
  the change of lipid marker, including Low-density lipoprotein cholesterol(LDL-C), total cholesterol(TC), High-density lipoprotein cholesterol(HDL-C), triglyceride(TG), non-HDL-C, between Rosuvastatin 10 mg/day and 20 mg/day treatment at 30 days.
the change of hsCRP | 30 days
  The change of inflammatory marker High sensitivity C-reactive protein(hsCRP) between Rosuvastatin 10 mg/day and 20 mg/day treatment at 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, M.D., Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Yeh RW, Sidney S, Chandra M, Sorel M, Selby JV, Go AS. Population trends in the incidence and outcomes of acute myocardial infarction. N Engl J Med. 2010 Jun 10;362(23):2155-65. doi: 10.1056/NEJMoa0908610. PMID 20558366
- [Result] Pasceri V, Patti G, Nusca A, Pristipino C, Richichi G, Di Sciascio G; ARMYDA Investigators. Randomized trial of atorvastatin for reduction of myocardial damage during coronary intervention: results from the ARMYDA (Atorvastatin for Reduction of MYocardial Damage during Angioplasty) study. Circulation. 2004 Aug 10;110(6):674-8. doi: 10.1161/01.CIR.0000137828.06205.87. Epub 2004 Jul 26. PMID 15277322
- [Result] Winchester DE, Wen X, Xie L, Bavry AA. Evidence of pre-procedural statin therapy a meta-analysis of randomized trials. J Am Coll Cardiol. 2010 Sep 28;56(14):1099-109. doi: 10.1016/j.jacc.2010.04.023. Epub 2010 Aug 31. PMID 20825761
- [Result] Yun KH, Oh SK, Rhee SJ, Yoo NJ, Kim NH, Jeong JW. 12-month follow-up results of high dose rosuvastatin loading before percutaneous coronary intervention in patients with acute coronary syndrome. Int J Cardiol. 2011 Jan 7;146(1):68-72. doi: 10.1016/j.ijcard.2010.04.052. Epub 2010 May 14. PMID 20471117
- [Result] Yun KH, Jeong MH, Oh SK, Rhee SJ, Park EM, Lee EM, Yoo NJ, Kim NH, Ahn YK, Jeong JW. The beneficial effect of high loading dose of rosuvastatin before percutaneous coronary intervention in patients with acute coronary syndrome. Int J Cardiol. 2009 Nov 12;137(3):246-51. doi: 10.1016/j.ijcard.2008.06.055. Epub 2008 Aug 15. PMID 18706705
- [Result] Gao yuan et al. Comparison of Effects of Loading Dose Rosuvastatin VERSUS Atorvastatin Therapy in Non-ST Segment Elevation Acute Coronary Syndrome Patients. Journal of China Medical University. 2013; 42:235-239.